CLINICAL TRIAL: NCT07341828
Title: An Exploratory Clinical Study of Anti-CD20/B-cell Maturation Antigen(BCMA) Chimeric Antigen Receptor Autologous T Cell Product (C-CAR168) in the Treatment of Central Nervous System Autoimmune Diseases Refractory to Standard Therapy
Brief Title: A Study of C-CAR168 in the Treatment of Central Nervous System Autoimmune Diseases Refractory to Standard Therapy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Principal Investigator, Xiangjun Chen, Professor of Neurology, Huashan Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-1015
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis (MS); Neuromyelitis Optica Spectrum Disorders (NMOSD); Autoimmune Encephalitis; Stiff Person Syndrome
Keywords: CD20/BCMA-directed CAR-T cells
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; Autoimmune Diseases of the Nervous System; Stiff-Person Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-CAR168 (Experimental): Autologous C-CAR168 administered by intravenous (IV) infusion
  Interventions: Biological: CD20/BCMA-directed CAR-T cells

INTERVENTIONS:
Biological: CD20/BCMA-directed CAR-T cells — Autologous 2nd generation CD20/BCMA-directed CAR-T cells, single infusion intravenously
  Other Names: C-CAR168

SUMMARY:
This is an investigator-initiated, single-center, open-label study of C-CAR168, an autologous bi-specific CAR-T therapy targeting CD20 and BCMA, for the treatment of adult patients with central nervous system autoimmune diseases refractory to standard therapy

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old at the time of signing the Informed Consent Form (ICF).
* Diagnosed as Multiple Sclerosis (MS)/Neuromyelitis Optica Spectrum Disorders (NMOSD)/Autoimmune Encephalitis(AiE)/Stiff Person Spectrum Disorder(SPSD) according to recognized diagnostic criteria for at least 6 months.
* Prior treatment failure with standard therapy.
* Adequate bone marrow, coagulation, cardiopulmonary, liver and renal function.

Exclusion Criteria:

* Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV), Treponema Pallidum (TP) positive, Cytomegalovirus (CMV) DNA positive, Epstein-Barr Virus (EBV) DNA positive.
* Uncontrolled active infection.
* Live vaccine injection within 4 weeks prior to signing the ICF.
* Major organ transplantation history or bone marrow/hematopoietic stem cell transplantation history.
* Severe cardiovascular diseases within the past 6 months prior to screening.
* A history of ≥ Grade 2 bleeding within 4 weeks prior to screening, or requiring long-term anticoagulants treatment.
* Inadequate washing time for previous treatment.
* Previously treated with CAR-T cell products or genetically modified T cell therapies.
* Pregnant or lactating women.
* Severe central nervous system diseases or pathological changes.
* Malignancy history within 5 years prior to signing the ICF.
* Any contraindication to lumbar puncture.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events [Safety and Tolerability] | Throughout the first 3 months follow up period completion
  Incidence and severity of adverse events (AE) and serious adverse events (SAE) within three months following infusion
The subsequent recommended dose of C-CAR168 in patients with central nervous system autoimmune diseases refractory to standard therapy | Throughout the first 24 months follow up period completion
  Based on the assessment of overall safety profile

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AE) | Throughout the first 24 months follow up period completion
  Incidence and severity of adverse events (AE) and serious adverse events (SAE) during the study
MS: No Evidence of Disease Activity-3 (NEDA-3) | Throughout the first 24 months follow up period completion
  Proportion of participants achieving NEDA-3 at 6 months post-infusion and during the study period
MS and NMOSD: Expanded Disability Status Scale (EDSS) | Throughout the first 24 months follow up period completion
  Change from baseline in EDSS at 6 months and 24 months post-infusion. EDSS and its associated functional system (FS) score provide a system for quantifying disability and monitoring changes in the level of disability over time. EDSS consists of 7 FS (visual FS, brainstem FS, pyramidal FS, cerebellar FS, sensory FS, bowel and bladder FS, and cerebral FS) which are used to derive EDSS score ranging from 0 (normal neurological exam) to 10 (death).
MS and NMOSD: MRI | Throughout the first 24 months follow up period completion
  Number of T1 gadolinium-enhancing lesions and new or enlarging T2 lesions, as well as their change from baseline, at 6 months and 24 months post-infusion. Change from baseline in total T2 lesion volume, gray matter volume (GMV), white matter volume (WMV), and brain volume (BV), as well as annualized-brain volume loss (a-BVL), at 6 months and 24 months post-infusion
Autoimmune Encephalitis (AiE): Clinical Assessment Scale in Autoimmune Encephalitis (CASE) | Throughout the first 24 months follow up period completion
  Change from baseline in CASE at 6 months and 24 months post-infusion. The Clinical Assessment Scale in Autoimmune Encephalitis (CASE) has a score range from 0 to 27, and higher scores indicate a worse clinical outcome.
MS, NMOSD and AiE: Annualized Relapse Rate (ARR) | Throughout the first 24 months follow up period completion
  ARR at 6 months and 24 months post-infusion
Stiff-Person Syndrome (SPS): Distribution of Stiffness Index (DSI) | Throughout the first 24 months follow up period completion
  Change from baseline in DSI at 6 months and 24 months post-infusion. Distribution of Stiffness Index (DSI) is a validated indicator or stiffness. Scores range from 0 to 6 and reflect the extent of stiffness. Higher scores indicate a worse outcome.
SPS: Heightened Sensitivity Score (HSS) | Throughout the first 24 months follow up period completion
  Change from baseline in HSS at 6 months and 24 months post-infusion. Heightened Sensitivity Score (HSS) measures changes in the frequency of spasms. Scores range from 0 to 7. Higher scores indicate a worse outcome.
Pharmacokinetics (PK): Maximal plasma concentration (Cmax) | Throughout the first 24 months follow up period completion
  Cmax of C-CAR168 in peripheral blood
PK: Time to reach the maximal plasma concentration (Tmax) | Throughout the first 24 months follow up period completion
  Tmax of C-CAR168 in peripheral blood
PK: Duration in peripheral blood (Tlast) | Throughout the first 24 months follow up period completion
  Tlast of C-CAR168 in peripheral blood
PK: Area under curve (AUC) | Throughout the first 24 months follow up period completion
  AUC of C-CAR168 in peripheral blood
Pharmacodynamics (PD): Depletion of peripheral blood B cells, plasma cells, and CD20dim T cells | Throughout the first 24 months follow up period completion
PD: Decline of serum immunoglobulin | Throughout the first 24 months follow up period completion

OTHER OUTCOMES:
Serum cytokines changes | Throughout the first 24 months follow up period completion
  Detection of serum cytokines changes over time by flow cytometry
Soluble BCMA changes in peripheral blood | Throughout the first 24 months follow up period completion
  Detection of soluble BCMA changes in peripheral blood by Enzyme Linked ImmunoSorbent Assay (ELISA)
Changes in CSF CAR DNA copy number and CAR-T cells | Throughout the first 24 months follow up period completion
  Detection of changes in CSF CAR DNA copy number and CAR-T cells by quantitative polymerase chain reaction (qPCR) and flow cytometry

IPD SHARING:
Plan to Share IPD: No